CLINICAL TRIAL: NCT01780116
Title: An Evaluation of the Effectiveness of Adherence Therapy for Schizophrenia: A Randomized Controlled Trial
Brief Title: Effectiveness of Adherence Therapy for Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Castle Peak Hospital (Other Government); Kwai Chung Hospital (Other)
Responsible Party: Principal Investigator, Chien Wai-Tong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AT-2013
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: schizophrenia; adherence therapy; medication; randomized controlled trial; cost-effectiveness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medicaiton adherence therapy (Experimental): Adherence therapy, consisting of six, 2-hour sessions over 3 months, in three phases:
  1. Engaging patients: assessing needs and concerns in medication adherence;
  2. Reviewing strengths and barriers and developing coping strategies; and
  3. Rationalizing beliefs and concerns and preventing relapse.
  Interventions: Behavioral: Adherence therapy
- Routine community care (No Intervention): Routine Community psychiatric nursing services provided by the Community Psychiatric Nurses in the practice field

INTERVENTIONS:
Behavioral: Adherence therapy — Systematic and highly structured medication adherence program using the motivational interviewing (MI) technique that focuses on six principles: expressing empathy, developing discrepancy between client's beliefs and evidence, supporting self-efficacy, avoiding argumentation, and rolling with resistance to behavioral change. MI is often able (with in-depth behavioral analysis) to focus on particular consequences of problem behavior, such as medication non-adherence, that have an obvious impact on patients.
  Other Names: Medication adherence program
  Arms: Medicaiton adherence therapy

SUMMARY:
When compared with those in the control (usual care) group, participants in the AT group are expected to demonstrate significant improvements immediately and at three, six and 12 months after completion of the intervention in: level of medication adherence, readmission rate, mental status, insight into treatment, and level of functioning.

DETAILED DESCRIPTION:
When compared with those in the control (usual care) group, participants in the AT group are expected to demonstrate significant improvements immediately and at three, six and 12 months after completion of the intervention in the following aspects:

1. level of adherence to antipsychotic medication,
2. rate and length of psychiatric hospital readmission,
3. mental status,
4. insight and attitude into illness and treatment, and
5. level of functioning.

The primary outcomes are level of antipsychotic medication adherence, re-hospitalization rates and mental status; and the patients' drug attitude will be the mediating factor of the AT.

ELIGIBILITY:
Inclusion Criteria of the patients include those who:

* are Hong Kong Chinese residents;
* have a primary diagnosis of schizophrenia or its subtypes such as schizophreniform and schizoaffective disorders not more than 3 years;
* have been prescribed oral antipsychotics for at least 1 month;
* are aged 18-65 years;
* have Positive and Negative Syndrome Scale (PANSS) score >60 and are judged by the case Community Psychiatric Nurse/psychiatrist as non-adherents; and
* are able to understand Cantonese/Mandarin.

Patients will be excluded if they have:

* only depot/intramuscular injections as regular psychiatric medication;
* co-morbidity of learning disability and organic brain disease, or clinically significant medical diseases;
* participated in adherence therapy; and/or
* visual, language or communication difficulty.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
re-hospitalization rate | 12 months after completion of intervention
  rate and length of psychiatric hospital readmission immediately, 6 months and 12 months after the completion of the intervention undertaken

SECONDARY OUTCOMES:
level of medication adherence | 12 months follow-up
  level of adherence to antipsychotic medication measured at recruitment and at immediately, 6 months and 12 months after completion fo the intervention
mental status | 12 months follow-up
  symptom severity measured at recruitment and at immediately, 6 months and 12 months after completion fo the intervention
insight into treatment | 12 months follow-up
  insights into illness and treatment measured at recruitment and at immediately, 6 months and 12 months after completion fo the intervention
functioning | 12 months follow-up
  level of functioning measured at recruitment and at immediately, 6 months and 12 months after completion fo the intervention

OTHER OUTCOMES:
program attendance and attrition | 12 months follow-up
  attendance and attrition rate

CONTACTS AND LOCATIONS:
Overall Officials: WT Chien, PhD, Principal Investigator — The Hogn Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Kwai Chung Hospital, Kwai Chung, NT
  - Castle Peak Hospital, Tuenmen, NT

REFERENCES:
- [Background] Chien WT, Leung SF, Yeung FK, Wong WK. Current approaches to treatments for schizophrenia spectrum disorders, part II: psychosocial interventions and patient-focused perspectives in psychiatric care. Neuropsychiatr Dis Treat. 2013;9:1463-81. doi: 10.2147/NDT.S49263. Epub 2013 Sep 25. PMID 24109184
- [Result] Chien, W.T., Mui, J., Cheung, E., & Gray, R. (2013). Effectiveness of medication adherence therapy for schizophrenia: A randomized controlled trial. Presentation (Book of Abstracts, pp. 144-146) at the 19th International Network for Psychiatric Nursing Research, 'The Personal and Political of Mental Health Nursing Research' (5-6 September 2013), Warwick Conference Centre, Coventry, UK. London: Royal College of Nursing.
- [Result] Chien WT, Mui JH, Cheung EF, Gray R. Effects of motivational interviewing-based adherence therapy for schizophrenia spectrum disorders: a randomized controlled trial. Trials. 2015 Jun 14;16:270. doi: 10.1186/s13063-015-0785-z. PMID 26072311
- [Derived] Chien WT, Mui J, Gray R, Cheung E. Adherence therapy versus routine psychiatric care for people with schizophrenia spectrum disorders: a randomised controlled trial. BMC Psychiatry. 2016 Feb 25;16:42. doi: 10.1186/s12888-016-0744-6. PMID 26911397